CLINICAL TRIAL: NCT06331481
Title: The Effect of Over Weight on Oocytes Quality in IVF Patients
Acronym: IVF
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0005-22-HYMC
Record Dates: First submitted 2024-03-07; First posted 2024-03-26 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: IVF; Overweight
MeSH Terms: conditions — Overweight | interventions — Cytological Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fullicular fluid for cytology and biochemical analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Fullicular fluid for cytology and biocemical analysis — The fullicular fluid in the oocyte retrieval process is consider to medical waste. This fluid contains a verity of proteins, mitochondria and verity of cells.
  The investigators using this fluid to learn about the evironment of the oocyte and its quality.

SUMMARY:
Obesity is an increasing worldwide problem and a risk factor for many diseases. The effect of obesity on female fertility has been extensively tested. Obese women have increased time to pregnancy and remain subfertile even in the absence of ovulatory dysfunction. They present with higher incidence of infertility compared to normal weight women.

This study is prospective observational cohort study performed between February 2022 until June 2022 in a single university-affiliated hospital.

DETAILED DESCRIPTION:
The effect of obesity on female fertility has been extensively tested. Obese women have increased time to pregnancy and remain subfertile even in the absence of ovulatory dysfunction. They present with higher incidence of infertility compared to normal weight women. Furthermore, obesity affects the outcome of fertility treatments, resulting in decreased ovarian response to stimulation, lower quantity and quality of oocytes, and adverse effects on the quality of embryos including lower blastocyst formation and on the chances of conception.

Subfertility and infertility research are aiming to find different markers that may shed light about oocyte quality. It is known that follicular fluid is the microenvironment of the oocyte. Both cumulus cells (CCs) and follicular fluid (FF) are critical determinants for oocyte and reflect its quality.

The oocyte in the ovary develops with the support of cumulus and granulosa cells, which are in close contact with her by gap junction. The oocytes are known to be unable to synthesize their own cholesterol and have very poor glucose metabolism to produce energy. The oocytes are supported for this purpose by cumulus and granulosa cells, and they basically reflect the quality of the oocytes. Evaluating different markers in the follicular fluid and cumulus cells including mitochondrial-DNA and protein that are known to be biomarkers of quality may help us to understand the impact of obesity on oocyte quality without harming the valuable resource.

In this study, the investigators aimed to evaluate the impact of obesity on oocyte quality using 2 main factors reflecting oocyte quality mtDNA levels in CCs and levels of proteins BMP-15 and HSPG2 in FFs.

Women younger than age 41 years, undergoing IVF/IVF-ICSI cycles, participated in the study. Patients were allocated into two BMI groups (<25 and >30) based on WHO criteria to evaluate distinctly different groups. The attending physician determined each patient's care plan without any relation to study recruitment. At the time of ultrasound-guided transvaginal ovum pick-up (OPU), only patients with four or more follicles were recruited. Demographic information was recorded from the electronic medical records, including demographics and obstetrical history (age, parity, BMI, number of previous pregnancies and abortions, prior IVF/ICSI cycles, and biochemical and basal hormonal profile), cycle characteristics (the stimulation protocol, endometrial thickness, and E2, LH and progesterone levels on hCG administration day), cycle outcomes (fertilization rate, number of oocytes, transferred and frozen embryos) and treatment outcomes (chemical and clinical pregnancy rate). Women who had undergone fertility preservation or had comorbidities, such as endocrine disorders, cancer, or other chronic diseases, were excluded.

ELIGIBILITY:
Inclusion Criteria:

1. All women divided by BMI below 25 and above 25 who underwent IVF-ICSI treatment.
2. Consent to participate in the study.

Exclusion Criteria:

1. Patients older than 40 years
2. Fertility preservation
3. Unbalanced endocrine disorders
4. Less than 4 follicles at the time of oocyte pick-up

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — IVF patients who undergo oocyte retrieval
Study Population: IVF patients who undergo oocyte retrieval
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Impact of obesity on oocyte's mtDNA expression in Cumulus Cells | 6 months
  How obesity impacts oocyte quality through analysis of mtDNA expression in Cumulus Cells
Impact of obesity on oocyte quality through levels of protein BMP-15 | 6 months
  How obesity impacts oocyte quality through analysis of levels of protein BMP-15 in Follicular fluid.
Impact of obesity on oocyte quality through levels of protein HSPG2 | 6 months
  How obesity impacts oocyte quality through analysis of levels of protein HSPG2 in Follicular fluid.

SECONDARY OUTCOMES:
Impact of obesity on fertilization and pregnancy rates through analysis of mtDNA expression | 18 months
  How obesity impacts fertilization and pregnancy rates through analysis of mtDNA expression in Cumulus Cells
Impact of obesity on fertilization and pregnancy rates through levels of protein BMP-15 | 18 months
  How obesity impacts fertilization and pregnancy rates through analysis of levels of protein BMP-15 in Follicular fluid.
Impact of obesity on fertilization and pregnancy rates through levels of protein HSPG2 | 18 months
  How obesity impacts fertilization and pregnancy rates through analysis of levels of protein HSPG2 in Follicular fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Einat Shalom-Paz, p, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center - IVF Unit, Hadera, Israel